CLINICAL TRIAL: NCT06992713
Title: A Phase Ia, First-in-human, Clinical Study of the Safety, Tolerability, and Pharmacokinetics of H1710 for Injection in Participants With Advanced Solid Tumors
Brief Title: A Clinical Study Evaluating H1710 for Injection in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Hepalink Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H1710-002
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- H1710 for Injection (Experimental): Participants receive H1710 for Injection according to the protocol.
  Interventions: Drug: H1710 for Injection

INTERVENTIONS:
Drug: H1710 for Injection — Injection.
  Other Names: H1710

SUMMARY:
This is a phase Ia clinical study evaluating H1710 for Injection in Participants with advanced solid tumors.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of H1710 for Injection in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years≤ age ≤ 75 years, irrespective of gender, ethnicity, financial, and educational background.
* Signed Informed Consent Form (ICF) prior to screening.
* Participants with histologically or cytologically confirmed advanced solid tumors, who have failed standard treatment, or have no standard treatment, or intolerant to or not suitable for standard treatment.
* Participants must have measurable or evaluable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Predicted life expectancy of at least 3 months.
* Adequate bone marrow reserve and organ function within 7 days prior to first dose of H1710.

Exclusion Criteria:

* Presence of malignant tumor lesion(s) that is/are at high risk of bleeding as judged by the clinical study investigator.
* Active clinically significant bleeding or conditions with a high risk of hemorrhage.
* Major surgery or interventional therapy or significant trauma within 28 days prior to the first dose of H1710, or elective surgery during the clinical trial period.
* Spinal or epidural anesthesia or loco-regional anesthesia within 24 hours prior to the first dose of H1710.
* Primary brain tumors. Active brain/meningeal metastases or central nervous system involvement who have clinical symptoms requiring medical intervention within 28 days prior to the first dose of H1710.
* Poorly controlled pleural effusion, pericardial effusion or ascites requiring repeated drainage as determined by investigators to be unsuitable for inclusion.
* Any anti-tumor therapy within 28 days prior to first dose of H1710, except for those who can be included after judgment by investigators.
* Participants have another active invasive malignancy, except for those who can be included after judgment by investigators.
* Symptomatic congestive heart failure, unstable angina, sinus bradycardia, clinically uncontrollable hypertension, and ongoing cardiac arrhythmia.
* Uncontrolled diabetes as determined by investigators.
* History of clinically significant interstitial lung disease or pneumonia as determined by investigators.
* Participants have a history of myocardial infarction within 6 months or coronary stenting within 12 months or a history of arterial thromboembolic event within 3 months before the first dose of H1710.
* Participants received a live attenuated vaccine within 28 days before the first dose of H1710 and/or plan to receive live vaccines during the study period unless approved by the clinical investigator and Sponsor.
* Human immunodeficiency virus (HIV) infection or HIV positive, active Hepatitis B Virus (HBV) infection, active Hepatitis C Virus (HCV) infection. Except those who can be included after judgment by investigators.
* Participants who have active bacterial, fungal or viral (except hepatitis virus) infections within 14 days before the first dose of H1710 and require intravenous or oral administration of antibiotics and/or other anti-infective therapeutic drugs.
* Any adverse events due to prior anti-tumor therapy unresolved to ≤ Grade 1 of CTCAE 5.0 (except for toxicities judged by the clinical investigator to be of no safety risk, such as alopecia, other long term ≤ Grade 2 toxicities which would not impact the administration of H1710 and safety evaluation).
* Participation in a clinical study of biological drug within 28 days, or within 14 days or 5 half-lives for small-molecule agents, before first dose of H1710, or current participation in other therapeutic investigational clinical trials.
* Females who are pregnant or lactating or who intend to become pregnant during the clinical trial period and within 6 months after discontinuation of H1710 treatment. Female or Male who refuse using reliable birth control methods during the clinical trial period and within 6 months after discontinuation of H1710.
* Participants who have any clinically significant psychiatric, social, or medical condition that, as judged by the clinical investigator, could increase the subject's risk, interfere with protocol adherence, or affect the subject's ability to give informed consent are ineligible to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-09-04 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | Up to ~ 18 months
  Incidence and severity of adverse events, serious adverse events, according to NCI-CTCAE Version 5.0
Dose Limiting Toxicities（DLT） | Up to ~ 18 months
Maximum Tolerated Dose (MTD) | Up to ~ 18 months
Recommended Phase 2 Dose (RP2D) | Up to ~ 18 months

SECONDARY OUTCOMES:
Maximum Observed Concentration(Cmax) of H1710 | Up to ~ 18 months
  Blood samples will be collected to determine the Cmax of H1710.
Time of Maximum Concentration (Tmax)of H1710 | Up to ~ 18 months
  Time to reach H1710 maximum observed concentration
Area Under the Concentration (AUC) of H1710 | Up to ~ 18 months
  Blood samples will be collected to determine the AUC of H1710.
Terminal Half life( t½) of H1710 | Up to ~ 18 months
  Blood samples will be collected to determine the terminal half-life of H1710.
Clearance (CL) of H1710 | Up to ~ 18 months
  Blood samples will be collected to determine the CL of H1710.
Objective Response Rate (ORR) | Up to ~ 18 months
  Percentage of participants with best response of complete response (CR) or partial response (PR).
Disease Control Rate(DCR) | Up to ~ 18 months
  The proportion of participants with best overall response of complete response(CR) or partial response(PR) or disease stabilization(SD) after treatment.
Duration of Response (DOR) | Up to ~ 18 months]
  Time from complete response(CR) or partial response(PR) to objective disease progression or death to any cause.
Progression Free Survival (PFS) | Up to ~ 18 months
  The time from the start of the treatment until objective disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing
  - Peking University Shougang Hospital, Beijing
  - Shanghai East Hospital, Shanghai